CLINICAL TRIAL: NCT02295436
Title: Pharmacokinetics and Tolerability of Minodronic Acid Tablets in Healthy Chinese Subjects and Food and Age Effects on the Pharmacokinetics
Brief Title: Pharmacokinetics and Tolerability of Minodronic Acid and Food and Age Effects on the Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Weiyong Li, vice director of the pharmacy department, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: WHXH-MINO
Record Dates: First submitted 2014-11-12; First posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Osteoporosis
Keywords: minodronic acid; pharmacokinetics; tolerability; food; age; Chinese subjects
MeSH Terms: conditions — Osteoporosis | interventions — YM 529

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1-mg group (Experimental): Twelve healthy young subjects were administered a single oral dose of 1 mg minodronic acid tablets at day 1 and then received repeated oral doses of minodronic acid (1 mg) once daily for 7 days (day 3 to day 9).
  Interventions: Drug: minodronic acid
- 2-mg group (Experimental): Twelve healthy young subjects were administered a single oral dose of 2 mg minodronic acid tablets.
  Interventions: Drug: minodronic acid
- 4-mg group (Experimental): Twelve healthy young subjects were administered a single oral dose of 4 mg minodronic acid tablets under fasting state at period 1.After a washout period of 8 days, they received the same dosage under fed conditions (administrated 30 minutes before high-fat breakfast).
  Interventions: Drug: minodronic acid
- 1-mg elderly group (Experimental): Twelve healthy elderly subjects were administered a single oral dose of 1 mg minodronic acid tablets.
  Interventions: Drug: minodronic acid

INTERVENTIONS:
Drug: minodronic acid — comparison of different doses, ages and medication conditions
  Other Names: YM529/ONO-5920

SUMMARY:
The primary objective of the the study was to evaluate the pharmacokinetic properties of minodronic acid tablets following single and multiple oral administration in healthy Chinese subjects. Additionally, the effects of age and food on minodronic acid pharmacokinetics was also explored.

DETAILED DESCRIPTION:
This was a single-center, phase I study in healthy young (19-30 years) and elderly (60-65 years) volunteers, which was conducted in four parts. In Part 1, minodronic acid tablets were administered to young volunteers at doses of 1, 2, and 4 mg. In Part 2, after a single dose, young volunteers in the 1-mg dose group received repeated oral doses of minodronic acid once daily for 7 days. In Part 3, a single oral dose of minodronic acid 1 mg was administered to elderly volunteers. In part 4, after a washout period of 8 days, volunteers in the 4-mg dose group received a single dose of 4 mg minodronic acid under fed conditions (administrated 30 minutes before high-fat breakfast). Plasma samples were collected and plasma concentrations of minodronic acid were analyzed by LC-MS/MS. Tolerability was assessed throughout the study by physical examinations, vital signs measurement, laboratory analyses, and monitoring of adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were included based on the following criteria:

  * males or females aged 19 to 35 years for young subjects or aged 60 to 65 years for elderly subjects
  * body mass index between 19 and 24 kg/m2
  * thorax radiography and ECG with no abnormalities
  * normal blood pressure values
  * heart rate
  * laboratory test results (hematology, blood biochemistry, hepatic function, and urinalysis)
  * negative test results for HIV and hepatitis B.

Exclusion Criteria:

* Subjects were excluded if they had a heart disease or disorder
* A hepatic, renal, respiratory, immune system, or nervous system disorder
* Any of the following conditions:

  * pregnancy
  * breast-feeding
  * hypocalcemia
  * prescription or over-the-counter medication use (including herbal products) within 2 weeks before the initiation of the study
  * blood donation or participation in other clinical trials within 3 months before enrollment in the study
  * alcohol or drug abuse
  * smoking more than 10 a day
  * clinically significant allergies to drugs or foods
  * sitting blood pressure <80/50 mm Hg or >140/100 mm Hg
  * A ventricular rate <60 beats/min or >100 beats/min at rest.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Cmax | two months
  the maximum observed plasma concentration and
AUC | two months
  the area under the concentration-time curve

SECONDARY OUTCOMES:
adverse events | two months

CONTACTS AND LOCATIONS:
Overall Officials: Weiyong Li, PhD, Principal Investigator — Tongji Medical College, Huazhong University of Science and Technology

REFERENCES:
- [Derived] Zhou Y, He X, Li H, Ni Y, Xu M, Sattar H, Chen H, Li W. Pharmacokinetics and tolerability of minodronic acid tablets in healthy Chinese subjects and food and age effects on the pharmacokinetics. Clin Ther. 2015 Apr 1;37(4):869-76. doi: 10.1016/j.clinthera.2015.01.015. Epub 2015 Mar 5. PMID 25748293